CLINICAL TRIAL: NCT01548235
Title: A Multicentre, Open Label, Non-randomised, Non-interventional, Observational Safety Study in Subjects With Type 2 Diabetes Mellitus, Starting or Switching to NovoMix® 30 Treatment
Brief Title: Observational Safety Study in Subjects With Type 2 Diabetes Mellitus Starting or Switching to Biphasic Insulin Aspart 30 Treatment
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-1812
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BIAsp 30 users
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Prescribed biphasic insulin aspart 30 as part of routine care. Starting dose, dose titration and injection frequency determined individually by each physician.

SUMMARY:
This study is conducted in Europe. The aim of this study is to investigate safety and efficacy in subjects with type 2 diabetes mellitus starting or switching to biphasic insulin aspart 30 (NovoMix® 30) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who started insulin therapy with biphasic insulin aspart 30 and subjects who switched from other insulin regimens to biphasic insulin aspart 30 by prescription of their physician as part of routine clinical practice in order to improve glycemic control.
  The selection of patients was at the discretion of the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 423 (Actual)
Dates: Start 2006-02; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Incidence of SADR (serious adverse drug reactions) including major hypoglycaemia

SECONDARY OUTCOMES:
Change from baseline in HbA1c (glycosylated haemoglobin)
Mean FPG (fasting plasma glucose)
Overall, daytime and nocturnal frequency of hypoglycaemic events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Copenhagen S, Denmark

REFERENCES:
- [Result] Breum L, Almdal T, Eiken P, Lund P, Christiansen E; Danish BIAsp Study Group. Initiating or switching to biphasic insulin aspart 30/70 therapy in subjects with type 2 diabetes mellitus. An observational study. Rev Diabet Stud. 2008 Fall;5(3):154-62. doi: 10.1900/RDS.2008.5.154. Epub 2008 Nov 10. PMID 19099087
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com